CLINICAL TRIAL: NCT02044380
Title: An Open Label Trial of Afatinib in Treatment-naive or Chemotherapy Pre-treated Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring EGFR Mutation(s)
Brief Title: Afatinib in Patients With Non Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.48
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental): patient to receive a tablet containing 40 mg afatinib once a day, with the option to reduce the dose to 30 or 20 mg/day, based on individual tolerability
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 40, 30, or 20mg tablets taken once daily, dosage depending on tolerability

SUMMARY:
The main aim of this study is to evaluate the safety and tolerability of afatinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring Epidermal Growth Factor Receptor (EGFR) mutation(s) and have never been treated with an EGFR-Tyrosine Kinase Inhibitor (TKI)

ELIGIBILITY:
Inclusion criteria:

1. Locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC)
2. Epidermal Growth Factor Receptor (EGFR) mutation-positive results per the institution's testing methodology
3. Male or female patients age >=18 years
4. Adequate organ function, defined as all of the following:

   1. Absolute neutrophil count (ANC) >1500/mm3
   2. Platelet count>75,000/mm3
   3. Serum creatinine<1.5 times of the upper limit of (institutional) normal and/or creatinine clearance (measured or calculated)>45ml/min
   4. Total bilirubin <1.5 times upper limit of (institutional) normal
   5. Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) < three times the upper limit of (institutional) normal (if related to liver metastases < five times ULN)
5. Eastern Cooperative Oncology Group (ECOG) score between 0-2
6. Written informed consent by patient or guardian prior to admission into the trial that is consistent with International Conference on Harmonization (ICH)- Good Clinical Practice (GCP) guidelines and local law
7. Recovery from any previous therapy related toxicity to <=CTCAE Grade 1 at study entry (except for stable sensory neuropathy <=CTCAE Grade 2 and alopecia)

Exclusion criteria:

1. Prior treatment with an EGFR tyrosine kinase inhibitor (TKI)
2. Hormonal anti-cancer treatment within 2 weeks prior to start of trial treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted)
3. Radiotherapy within 28 days prior to drug administration, except as follows:

   1. Palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
   2. Single dose palliative treatment for symptomatic metastases outside above allowance to be discussed with sponsor prior to enrolling
4. Major surgery within 4 weeks before starting trial treatment or scheduled for surgery during the projected course of the trial
5. Known hypersensitivity to afatinib or any of its excipients
6. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to starting trial treatment
7. Women of Child-Bearing Potential (WOCBP) and men who are able to father a child, unwilling to use adequate contraception prior to trial entry, for the duration of trial participation and for at least 2 weeks after treatment has ended
8. Childbearing potential who:

   1. are nursing or
   2. are pregnant or
   3. are not using an acceptable method of birth control, or do not plan to continue using this method throughout the trial and/or do not agree to submit to pregnancy testing required by this protocol
9. Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patients ability to comply with the trial or interfere with the evaluation of safety for the trial drug
10. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured
11. Requiring treatment with any of the prohibited concomitant medications that cannot be stopped for the duration of trial participation
12. Known pre-existing interstitial lung disease
13. Presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug (e.g. Crohn's disease, ulcerative colitis, malabsorption, or Common Terminology Criteria grade =2 diarrhea of any aetiology) based on investigator assessment
14. Active hepatitis B infection (defined as presence of Hepatitis B (HepB) sAg and/or HepB DNA), active Hepatitis C (HEP C) infection (defined as presence of Hep C RNA) and/or known Human Immunodeficiency Virus (HIV) carrier
15. Meningeal carcinomatosis
16. Symptomatic brain metastases (patients with asymptomatic brain metastases, who were previously treated, are eligible provided they have had Stable Disease (SD) for at least 4 weeks on stable doses of corticosteroid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Canada (5):
  - Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, multicenter, single-arm trial evaluated the safety & tolerability of the investigational drug afatinib.All entered patients in this trial (i.e., patients that had been treated with the trial medication) received continuous treatment of afatinib in the absence of disease progression or meeting any other trial withdrawal criteria.
Pre-assignment Details: The planned trial end date was 10 February 2016. On the end date, all patients on treatment that met the approved label indication were planned to be switched to commercially available afatinib.
Groups:
- Afatinib 40 mg: Patient to receive a film coated tablet containing 40 mg afatinib once a day, with the option to reduce the dose to 30 or 20 mg/day, based on individual tolerability.
Period: Overall Study
Arm/Group | Afatinib 40 mg
Started | 14 (Started are the treated patients)
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set: This analysis set included all patients who were dispensed trial treatment (afatinib) and were documented to have taken at least one dose of afatinib.
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety Assesment
Description: Safety was assessed by:
  1. All serious adverse events (SAEs)
  2. All adverse events (AEs) leading to treatment discontinuation or dose reduction of afatinib
  3. Non-serious AEs assessed by the treating physician as related to afatinib.
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 80 weeks.
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 14
Percentage of participants
  Investigator defined drug-related AEs | 92.9
  AEs leading to dose reduction | 35.7
  AEs leading to discont. of trial drug | 35.7
  Serious AEs | 21.4

ADVERSE EVENTS:
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 80 weeks.
Arm/Group | Afatinib 40 mg
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=14)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 1
Radiation associated pain (Injury, poisoning and procedural complications) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=14)
Tachycardia (Cardiac disorders) | 1
Growth of eyelashes (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oesophagitis (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Body tinea (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Omphalitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 5
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Muscle spasticity (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Mood altered (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Scab (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the small number of patients entered and treated in this trial (14 patients) relative to the planned enrollment goal (40 entered patients had been planned), no formal statistical analyses of efficacy data were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.